CLINICAL TRIAL: NCT07171411
Title: The Combined Effects of Whey Protein and Collagen Supplementation on Bone Mineral Density and Muscle Mass in Resistance-Trained Men: A Randomized Controlled Trial
Brief Title: Combined Whey Protein and Collagen Supplementation in Resistance-Trained Men
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara Yildirim Beyazıt University (Other)
Collaborators: Saglik Bilimleri Universitesi (Other); Islamic Azad University of Mashhad (Other); Manisa Celal Bayar University (Other); Muş Alparslan University (Other); Pamukkale University (Other); Australian Catholic University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IAU.Ilk.C.162911421.2024
Record Dates: First submitted 2025-09-06; First posted 2025-09-12 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Muscle Hypertrophy; Bone Mineral Density Loss; Resistance Training Adaptation
Keywords: Whey Protein; Collagen Peptides; Resistance Training; Muscle Mass; Bone Mineral Density; Bone Turnover Biomarkers; Strength Training; Protein Supplementation; Hypertrophy; Sports Nutrition
MeSH Terms: conditions — Hypertrophy | interventions — Whey Proteins; Collagen; maltodextrin

STUDY DESIGN:
Intervention Model Description: Participants were randomly assigned into one of four parallel groups (Whey + Collagen, Whey only, Collagen only, Placebo). Each group received its allocated supplementation daily for 8 weeks in combination with a standardized resistance training program. Groups were followed concurrently with no crossover.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blind design extended to all relevant parties. Supplements were provided in identical, opaque sachets to ensure concealment. Randomization sequence was managed by an independent statistician not involved in data collection or analysis. Participants, trainers, investigators, and outcome assessors remained blinded to group assignments until completion of analyses.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Whey Protein + Collagen (WP+C) (Experimental): Participants received 30 g/day whey protein isolate plus 10 g/day type I & III collagen peptides, split into two daily doses (morning and post-exercise or at same time on rest days). Supplements were packaged in identical sachets.
  Interventions: Dietary Supplement: Whey Protein + Collagen
- Whey Protein Only (WP) (Active Comparator): Participants received 30 g/day whey protein isolate, split into two daily doses. Packaged identically to other interventions to maintain blinding.
  Interventions: Dietary Supplement: Whey Protein
- Collagen Only (C) (Active Comparator): Participants received 10 g/day type I & III collagen peptides, split into two daily doses. Identical packaging ensured blinding.
  Interventions: Dietary Supplement: Collagen Peptides
- Placebo (P) (Placebo Comparator): Participants received 10 g/day maltodextrin (isocaloric with protein groups), provided in identical sachets to ensure blinding.
  Interventions: Other: Maltodextrin (Placebo)

INTERVENTIONS:
Dietary Supplement: Whey Protein + Collagen — Participants consumed 30 g/day whey protein isolate (Optimum Nutrition) combined with 10 g/day type I & III collagen peptides (Vital Proteins). Supplements were provided as single-dose sachets, identical in appearance, and taken twice daily (morning and post-exercise or same time on rest days) for 8 weeks.
  Arms: Whey Protein + Collagen (WP+C)
Dietary Supplement: Whey Protein — Participants consumed 30 g/day whey protein isolate (Optimum Nutrition), in identical sachets, taken twice daily for 8 weeks.
  Arms: Whey Protein Only (WP)
Dietary Supplement: Collagen Peptides — Participants consumed 10 g/day type I & III collagen peptides (Vital Proteins), in identical sachets, taken twice daily for 8 weeks.
  Arms: Collagen Only (C)
Other: Maltodextrin (Placebo) — Participants consumed 10 g/day maltodextrin powder (isocaloric to protein supplements), packaged identically, taken twice daily for 8 weeks.
  Arms: Placebo (P)

SUMMARY:
This study tested whether taking whey protein together with collagen peptides would provide greater benefits for muscle and bone health compared to whey protein alone, collagen alone, or a placebo. Forty healthy, resistance-trained men aged 18-35 years were randomly assigned to one of four groups: (1) whey protein plus collagen (30 g + 10 g/day), (2) whey protein only (30 g/day), (3) collagen only (10 g/day), or (4) placebo (maltodextrin). All participants followed a supervised resistance training program (3 times per week) for 8 weeks.

The primary outcome was muscle mass, measured with bioelectrical impedance analysis (BIA). Secondary outcomes included bone mineral density (DXA scans), maximal strength (1RM squat and bench press), and blood markers of bone turnover (P1NP and CTX-I).

Results showed that the whey + collagen group achieved the largest improvements in muscle growth, lumbar spine bone mineral density, strength, and favorable changes in bone turnover markers compared to all other groups. No serious side effects were reported, and supplement adherence was very high.

These findings suggest that combining whey protein and collagen may be a practical strategy to support muscle and bone adaptation in resistance-trained men.

DETAILED DESCRIPTION:
This was a double-blind, randomized, placebo-controlled trial evaluating the combined effects of whey protein and collagen supplementation on muscle mass, bone mineral density (BMD), muscular strength, and bone turnover markers in resistance-trained men.

Forty healthy male participants (18-35 years, with ≥1 year of resistance training experience) were recruited and randomized into four parallel groups (n=10 per group):

Whey Protein + Collagen (30 g WP + 10 g collagen/day)

Whey Protein only (30 g/day)

Collagen only (10 g/day)

Placebo (10 g maltodextrin/day, isocaloric)

All supplements were provided in identical single-dose sachets to ensure blinding. Participants consumed one dose upon waking and one post-exercise (or same time on rest days). A standardized, supervised hypertrophy-oriented resistance training program (3 sessions/week for 8 weeks) was applied to all groups.

Primary outcome: Muscle mass (lean body mass, assessed with BIA at baseline and 8 weeks).

Secondary outcomes: Lumbar spine and femoral neck BMD (DXA), maximal squat and bench press strength (1RM), and serum biomarkers of bone turnover (P1NP and CTX-I).

The trial was approved by the Islamic Azad University IRB (Protocol No: IAU.Ilk.C.162911421.2024). All participants gave written informed consent. Compliance with supplementation was >90% and training adherence was >95%. No adverse events were reported.

ELIGIBILITY:
Inclusion Criteria:

* Male participants aged 18-35 years
* At least 1 year of consistent resistance training experience (≥3 sessions per week, targeting major muscle groups)
* Healthy, with no history of musculoskeletal, metabolic, or cardiovascular disorders
* No current or recent (<6 months) use of anabolic steroids, growth hormones, or performance-enhancing substances
* Non-smoker and no habitual use of anti-inflammatory medications
* Able and willing to comply with supplementation and supervised training program
* Provided written informed consent

Exclusion Criteria:

* Participation in similar supplementation studies in the past 6 months
* Recent fractures or surgeries affecting musculoskeletal health (<6 months)
* Known allergy or intolerance to dairy proteins or collagen supplements
* Inability to attend scheduled supervised resistance training sessions
* Non-adherence to dietary control requirements (e.g., use of additional protein/creatine supplements during study)
* Any condition deemed by investigators to interfere with study compliance or safety

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2024-01-03 (Actual); Primary Completion 2024-03-10 (Actual); Study Completion 2024-04-10 (Actual)

PRIMARY OUTCOMES:
Change in Muscle Mass (kg, lean body mass by BIA) | Baseline (week 0) to 8 weeks post-intervention
  Muscle mass was assessed using bioelectrical impedance analysis (InBody 770). Measurements were conducted under standardized conditions (≥8 h fasted, no exercise or caffeine for ≥12 h, urine specific gravity <1.020). Values reported as lean body mass (kg). Primary analysis compared changes between Whey + Collagen, Whey only, Collagen only, and Placebo groups after 8 weeks of supplementation combined with resistance training.

SECONDARY OUTCOMES:
Change in Lumbar Spine Bone Mineral Density (BMD) | Baseline to 8 weeks
  BMD measured at lumbar spine (L1-L4) using DXA (Hologic Discovery A). Scans performed by trained technician with daily calibration.
Change in Femoral Neck Bone Mineral Density (BMD) | Baseline to 8 weeks
  BMD measured at femoral neck using DXA, reported in g/cm².
Change in Squat Strength (1RM) | Baseline to 8 weeks
  Maximal squat strength (kg) assessed via 1-repetition maximum (1RM) testing under standardized protocol, supervised by certified trainers.
Change in Bench Press Strength (1RM) | Baseline to 8 weeks
  Maximal bench press strength (kg) assessed via standardized 1RM testing, supervised by certified trainers.
Change in Procollagen Type I N-Terminal Propeptide (P1NP) | Baseline to 8 weeks
  Serum P1NP, a marker of bone formation, measured via ELISA. Blood collected after overnight fast (7:00-9:00 AM), samples stored at -80°C.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Health Sciences, Ankara, Etlik, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) that support the findings of this study will be made available to qualified researchers upon reasonable request from the corresponding author. Requests will require approval by the Islamic Azad University Institutional Review Board to ensure compliance with ethical and data protection regulations. Supporting documents such as the study protocol and statistical analysis plan will also be available. Data will be shared beginning 6 months after publication of the study results and remain accessible for 5 years.
Supporting Information: Study Protocol, SAP
Time Frame: De-identified IPD, study protocol, and statistical analysis plan will be available starting 6 months after publication of the trial results. Data will remain available for a period of 5 years thereafter.
Access Criteria: Qualified academic and clinical researchers may request access to de-identified participant data, along with the study protocol and statistical analysis plan. Requests must be submitted in writing to the corresponding author and will be reviewed by the research team in consultation with the Institutional Review Board. Access will be granted for scientifically valid proposals. Data will be shared through secure transfer methods in compliance with data protection regulations.
URL: https://orcid.org/0000-0002-1524-6295